CLINICAL TRIAL: NCT00359372
Title: Predicting Response to Cardiac Resynchronization Therapy in Heart Failure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060216; 06-H-0216
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-29

CONDITIONS: Heart Failure; Left Ventricular Dysfunction
Keywords: Chronic Heart Failure; Cardiac Resynchronization; Magnetic Resonance Imaging; Biventricular Pacing; Heart Function; CRT
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

SUMMARY:
This study will explore which characteristics of patients with heart failure will likely predict improvement after cardiac resynchronization (CRT), implantation of a pacemaker to improve heart function. In spite of major medical advances, about 30% to 40% of patients with heart failure do not respond to CRT, and the reasons are not well understood. This study will involve magnetic resonance imaging (MRI), electrocardiogram (ECG), and echocardiography techniques to let researchers examine what may influence response to CRT.

Patients ages 18 and older with a left ventricular disorder and who are not pregnant or breastfeeding may be eligible for this study. Initial evaluation will take 5 to 6 hours. A blood sample of about 2 tablespoons will be collected, and several procedures will be performed. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. For that procedure, patients will lie on a table that slides into the enclosed tunnel of the scanner and be asked to lie still. They will be in the scanner for 30 to 90 minutes. As the scanner takes pictures, patients will hear knocking sounds, and they may be asked to hold their breath intermittently for 5 to 20 seconds. During part of the scan, a drug called gadolinium will be given intravenously (IV), to make the heart easier to see. Patients will be able to communicate with the MRI staff at all times during the scan. At any time, patients may ask to be moved out of the machine. Patients having metal in their body that interferes with the MRI scanner should not have this test. During the procedure, an ECG machine will monitor the heart, through wires connected to pads on the skin. Patients will have an echocardiogram, in which sound waves look at the heart. A small handheld probe will touch the chest and abdomen, and an IV tube may be inserted to inject a contrast drug to improve the quality of heart images. Patients will have a cardiopulmonary stress test (treadmill test) and a 6-minute walk test, both before pacemaker implantation and then 6 months afterward. Also before and after pacemaker implantation, patients will complete the Minnesota Living with Heart Failure Questionnaire, regarding the impact of heart failure on patients' lives. The follow-up visit will take 3 to 4 hours.

DETAILED DESCRIPTION:
Many patients with heart failure benefit from cardiac resynchronization therapy (CRT) which involves implantation of a pacemaker to improve the coordination of heart function. However, approximately 30-40% of patients fail to respond to this therapy with current selection criteria. We hypothesize that patients with echocardiographic and MRI measures of a high degree of LV mechanical dyssynchrony are more likely to benefit from CRT than patients with less baseline dyssynchrony. Severe LV remodeling as measured by MRI may also predict patients less likely to benefit from therapy. In addition, myocardial fibrosis/scarring as measured by MRI delayed enhancement imaging may predict segments or subjects less likely to respond to CRT even in patients without ischemic heart disease. In this study, patients with New York Heart Association class III - IV heart failure will undergo imaging and stress testing prior to CRT pacemaker implantation and 6 months later to determine predictors of response. Considering the complexity of the protocol and novelty of some aspects of the MRI examination, we consider this an exploratory observational protocol.

ELIGIBILITY:
* INCLUSION and EXCLUSION CRITERIA

No one will be excluded from this study based on race, gender, and ethnicity.

INCLUSION CRITERIA

1. LV dysfunction with an LV ejection fraction less than or equal to 35% (by clinical echocardiography, cardiac catheterization, radionuclide ventriculography, or MRI).
2. New York Heart Association (NYHA) class III or IV functional status
3. QRS interval greater than or equal to 120msec (measured on clinical ECG)
4. Optimal pharmacological therapy for heart failure with at least 1 month on an ACE-inhibitor or angiotensin II receptor blocker (ARB) and if on a beta blocker, 3 months on a stable dose of a beta blocker. Patients need to be taking their medicines consistently to be enrolled in this study.

EXCLUSION CRITERIA

1. Coronary artery bypass graft surgery or percutaneous coronary intervention within 60 days of enrollment.
2. Chronic medically refractory atrial tachyarrhythmias
3. History of medical non-compliance
4. Women who are pregnant or not using medically acceptable birth control (since the x-rays used to guide pacemaker therapy may increase the risk to the fetus and the fetal risks of gadolinium are not well known).
5. Contraindication to MRI scanning including patients with the following devices:

   i. Central nervous system aneurysm clips

   ii. Implanted neural stimulator

   iii. Implanted cardiac pacemaker or defibrillator prior to enrollment

   iv. Cochlear implant

   v. Ocular foreign body (e.g. metal shavings)

   vi. Insulin pump

   vii. Metal shrapnel or bullet
6. Contraindications to MRI contrast agent administration:

   i. lactating women

   ii. patients with hemoglobinopathies

   iii. severe renal disease (CrCl less than 20 ml/min)
7. Baseline 6-minute hall walk distance more than 450 meters (to exclude patients who are unlikely to truly have NYHA class III to IV heart failure)
8. Enrollment in any concurrent study that may confound the results of this study
9. Life expectancy less than 6 months because of other medical conditions.
10. Age less than 18 years since this disease is not prevalent in children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2006-07-28; Study Completion 2007-05-29

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mid-Atlantic Associates, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368